CLINICAL TRIAL: NCT06734650
Title: Development and Validation of a Peripheral Venous Waveform-based Pulse Pressure Variation Calculating Deep Learning Model
Brief Title: Deep Learning Model for Predicting a Peripheral Venous Waveform-based Pulse Pressure Variation
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Park InSun, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2411-936-303
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Vein; Arterial Wave Reflections; Pulse Pressure Variation; Stroke Volume Variation; Deep Learning Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral waveform collection group: 1. Peripheral Venous Pressure Variation
  2. Stroke Volume Variation
  3. Pulse Pressure Variation
  4. Pleth Variability Index
  Interventions: Other: peripheral waveform collection

INTERVENTIONS:
Other: peripheral waveform collection — The peripheral venous pressure waveform is collected by connecting a pressure transducer that is currently in use to the placed central venous line. In addition, the pulse pressure variation or stroke volume variation value that can be obtained from the arterial catheter. This extracts the medical records and bio-signal information of the subjects registered through the previously approved 'Establishment of a Bio-signal and Clinical Information Registry for the Development of Patient Monitoring Algorithm' study (B-2202-738-401).

SUMMARY:
Pulse pressure variation is a monitoring index that indicates the response to fluid therapy in patients receiving mechanical ventilation, and is used as a reference for patients with unstable hemodynamic conditions. However, it is invasive because it requires arterial puncture to collect it. In a previous study by the investigators, the investigators developed and verified an artificial intelligence model that predicts stroke volume variation, in real time using only the central venous pressure waveform. However, since a large vein such as the jugular vein must be punctured to collect the central venous pressure waveform, it is still invasive, and its clinical utility is low. Therefore, in this study, the investigators collected waveforms from peripheral veins that are less invasive and can be a wide range of applications because all surgical patients have them. The investigators aimed to develop and verify an artificial intelligence model that predicts pulse pressure variation obtained from peripheral venous waveforms .

DETAILED DESCRIPTION:
In this study, the investigators collected waveforms from peripheral veins that are less invasive and can be a wide range of applications because all surgical patients have them. The investigators aimed to develop and verify an artificial intelligence model that predicts pulse pressure variation obtained from peripheral venous waveforms .

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily agreed and signed the written informed consent form before participating in this study
* Adult aged 19 years or older
* American Society of Anesthesiologists physical class (ASA) 1-3
* Patients scheduled for elective hepatectomy under general anesthesia
* Patients who require arterial pressure monitoring and additional peripheral venous access for routine anesthesia preparation
* Non-smokers with normal pulmonary function

Exclusion Criteria:

* Patients with abnormal findings on electrocardiogram before surgery
* Patients who cannot undergo peripheral venous puncture

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective hepatectomy under general anesthesia
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Pulse pressure variation | intraoperative period
  from arterial waveform

CONTACTS AND LOCATIONS:
Overall Officials: Insun Park, M.D./Ph.D., Principal Investigator — assistant professor
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyunggi-do, South Korea